CLINICAL TRIAL: NCT04330638
Title: A Prospective, Randomized, Factorial Design, Interventional Study to Compare the Safety and Efficacy of Combinations of Blockade of Interleukin-6 Pathway and Interleukin-1 Pathway to Best Standard of Care in Improving Oxygenation and Short- and Long-term Outcome of COVID-19 Patients With Acute Hypoxic Respiratory Failure and Systemic Cytokine Release Syndrome
Brief Title: Treatment of COVID-19 Patients With Anti-interleukin Drugs
Acronym: COV-AID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Belgium Health Care Knowledge Centre (Other Government)
Responsible Party: Principal Investigator, Bart N. Lambrecht, Professor in Pulmonology, Director VIB-Inflammational Research Center, University Hospital, Ghent
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: COV-AID
Record Dates: First submitted 2020-03-31; First posted 2020-04-01 (Actual); Results first posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
Keywords: Acute Lung Injury; Hypoxia; Acute Respiratory Distress Syndrome; Corona virus; COVID-19; SARS (Severe Acute Respiratory Syndrome); Systemic Cytokine release Syndrome
MeSH Terms: conditions — COVID-19; Acute Lung Injury; Hypoxia; Respiratory Distress Syndrome; Severe Acute Respiratory Syndrome | interventions — Interleukin 1 Receptor Antagonist Protein; siltuximab; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Usual Care (Placebo Comparator)
  Interventions: Other: Usual Care
- Anakinra (Active Comparator)
  Interventions: Drug: Anakinra
- Siltuximab (Active Comparator)
  Interventions: Drug: Siltuximab
- Anakinra + Siltuximab (Active Comparator)
  Interventions: Drug: Anakinra; Drug: Siltuximab
- Tocilizumab (Active Comparator)
  Interventions: Drug: Tocilizumab
- Anakinra + Tocilizumab (Active Comparator)
  Interventions: Drug: Anakinra; Drug: Tocilizumab

INTERVENTIONS:
Other: Usual Care — Usual Care
  Arms: Usual Care
Drug: Anakinra — Anakinra will be given as a daily subcutaneous injection of 100 mg for 28 days or until hospital discharge, whichever is first
  Other Names: KINERET®
  Arms: Anakinra; Anakinra + Siltuximab; Anakinra + Tocilizumab
Drug: Siltuximab — Siltuximab will be given via single IV infusion at a dose of 11 mg/kg
  Other Names: SYLVANT®
  Arms: Anakinra + Siltuximab; Siltuximab
Drug: Tocilizumab — Tocilizumab will be given via single IV infusion at a dose of 8 mg/kg with a maximum infusion of 800 mg/injection
  Other Names: ROACTEMRA®
  Arms: Anakinra + Tocilizumab; Tocilizumab

SUMMARY:
The purpose of this study is to test the safety and effectiveness of individually or simultaneously blocking IL-6 and IL-1 versus standard of care on blood oxygenation and systemic cytokine release syndrome in patients with COVID-19 coronavirus infection and acute hypoxic respiratory failure and systemic cytokine release syndrome

DETAILED DESCRIPTION:
There are currently no treatments directed at halting the cytokine storm and acute lung injury to stop the progression from manageable hypoxia to frank respiratory failure and ARDS in patients with COVID-19 infection. Preventing progression from early acute hypoxia and cytokine release syndrome to frank hypoxic respiratory failure and ARDS could have a huge impact on the foreseeable overflow of the ICU units. In ventilated patients, preventing the onset of ARDS, or shortening ICU stay could also be crucial in this regard.

The clinical status after 15 days treatment is evaluated to measure the effectiveness of tocilizumab, tocilizumab and anakinra, siltuximab, siltuximab and anakinra and anakinra on restoring lung homeostasis,using single IV injection (siltuximab or tocilizumab) combined or not with daily subcutaneous injections of anakinra until 28 days or hospital discharge, whichever is first. During the treatment period, daily clinical assesments of severity, daily laboratory check-up, measurements of oxygen saturation (pulse oximetry) in relation to FiO2, regular arterial blood gas measurements, regular chest X-rays, chest CT scans on indication will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Recent ( ≥ 6 days of flu-like symptoms or malaise yet ≤16 days of flu-like symptoms or malaise prior to randomization) infection with COVID-19.
* Confident COVID-19 diagnosis confirmed by antigen detection test and/or PCR and/or positive serology, or any emerging and validated diagnostic laboratory test for COVID-19 within this period.
* In some patients, it may be impossible to get a confident laboratory confirmation of COVID-19 diagnosis after 24h of hospital admission because viral load is low and/or problems with diagnostic sensitivity. In those cases, in absence of an alternative diagnosis, and with highly suspect bilateral ground glass opacities on recent (<24h) chest-CT scan (confirmed by a radiologist and pulmonary physician as probable COVID-19), and a typical clinical and chemical diagnosis with signs of cytokine release syndrome, a patient can be enrolled as probable COVID-19 infected. In all cases, this needs confirmation by later seroconversion.
* Presence of hypoxia defined as PaO2/FiO2 below 350 while breathing room air in upright position or PaO2/FiO2 below 280 on supplemental oxygen and immediately requiring high flow oxygen device or mechanical ventilation
* signs of cytokine release syndrome defined as ANY of the following:

  1. serum ferritin concentration >1000 mcg/L and rising since last 24h
  2. single ferritin above 2000 mcg/L in patients requiring immediate high flow oxygen device or mechanical ventilation
  3. lymphopenia defined as <800 lymphocytes/microliter) and two of the following extra criteria

     * Ferritin > 700 mcg/L and rising since last 24h
     * increased LDH (above 300 IU/L) and rising last 24h
     * D-Dimers > 1000 ng/mL and rising since last 24h
     * CRP above 70mg/L and rising since last 24h and absence of bacterial infection
     * if three of the above are present at admission, no need to document 24h rise
* Chest X-ray or CT scan showing bilateral infiltrates within last 2 days
* Admitted to specialized COVID-19 ward or an ICU ward taking care of COVID-19 patients
* Age ≥ 18yrs
* Male or Female
* Willing and able to provide informed consent or legal representative willing to provide informed consent

Exclusion Criteria:

* Patients with known history of serious allergic reactions, including anaphylaxis, to any of the study medications, or any component of the product.
* mechanical ventilation > 24 h at Randomization
* Patient on ECMO at time of screening
* clinical frailty scale above 3 (This frailty score is the patient status before first symptoms of COVID-19 episode.)
* active bacterial or fungal infection
* unlikely to survive beyond 48h
* neutrophil count below 1500 cells/microliter
* platelets below 50.000/microliter
* Patients enrolled in another investigational drug study
* patients on high dose systemic steroids (> 20 mg methylprednisolone or equivalent) for COVID-19 unrelated disorder
* patients on immunosuppressant or immunomodulatory drugs
* patients on current anti-IL1 or anti-IL6 treatment
* signs of active tuberculosis
* serum transaminase levels >5 times upper limit of normal
* bowel perforation or diverticulitis
* pregnant or breastfeeding females (all female subjects deemed of childbearing potential by the investigator must have negative pregnancy test at screening)
* Women of childbearing potential must have a negative serum pregnancy test pre-dose on day 1. Woùmen of childbearing potential must consistently and correctly use (during the entire treatment period and 3 months after last reatment) 1 highly effective method for contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Lambrecht, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (15):
- Belgium (15):
  - AZ Sint-Jan Brugge, Bruges
  - University Hospital Saint-Pierre, Brussels
  - Erasmus University Hospital, Brussels
  - University Hospital Saint-Luc, Brussels
  - University Hospital Antwerp, Edegem
  - Ziekenhuis Oost-Limurg, Genk
  - AZ Sint-Lucas, Ghent
  - University Hospital Ghent, Ghent
  - Jessa ZH, Hasselt
  - University Hospital Brussels, Jette
  - CHU Tivoli, La Louvière
  - CHR de la Citadelle, Liège
  - University Hospital Liège, Liège
  - Cliniques Saint-Pierre Ottignies, Ottignies-Louvain-la-Neuve
  - AZ Delta, Roeselare

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Davidson M, Menon S, Chaimani A, Evrenoglou T, Ghosn L, Grana C, Henschke N, Cogo E, Villanueva G, Ferrand G, Riveros C, Bonnet H, Kapp P, Moran C, Devane D, Meerpohl JJ, Rada G, Hrobjartsson A, Grasselli G, Tovey D, Ravaud P, Boutron I. Interleukin-1 blocking agents for treating COVID-19. Cochrane Database Syst Rev. 2022 Jan 26;1(1):CD015308. doi: 10.1002/14651858.CD015308. PMID 35080773
- [Derived] Declercq J, Van Damme KFA, De Leeuw E, Maes B, Bosteels C, Tavernier SJ, De Buyser S, Colman R, Hites M, Verschelden G, Fivez T, Moerman F, Demedts IK, Dauby N, De Schryver N, Govaerts E, Vandecasteele SJ, Van Laethem J, Anguille S, van der Hilst J, Misset B, Slabbynck H, Wittebole X, Lienart F, Legrand C, Buyse M, Stevens D, Bauters F, Seys LJM, Aegerter H, Smole U, Bosteels V, Hoste L, Naesens L, Haerynck F, Vandekerckhove L, Depuydt P, van Braeckel E, Rottey S, Peene I, Van Der Straeten C, Hulstaert F, Lambrecht BN. Effect of anti-interleukin drugs in patients with COVID-19 and signs of cytokine release syndrome (COV-AID): a factorial, randomised, controlled trial. Lancet Respir Med. 2021 Dec;9(12):1427-1438. doi: 10.1016/S2213-2600(21)00377-5. Epub 2021 Oct 29. PMID 34756178
- [Derived] Brands X, de Vries FMC, Uhel F, Haak BW, Peters-Sengers H, Schuurman AR, van Engelen TSR, Lutter R, Cremer OL, Bonten MJ, Schultz MJ, Scicluna BP, van der Poll T; MARS Consortium. Plasma Ferritin as Marker of Macrophage Activation-Like Syndrome in Critically Ill Patients With Community-Acquired Pneumonia. Crit Care Med. 2021 Nov 1;49(11):1901-1911. doi: 10.1097/CCM.0000000000005072. PMID 33935163
- [Derived] Maes B, Bosteels C, De Leeuw E, Declercq J, Van Damme K, Delporte A, Demeyere B, Vermeersch S, Vuylsteke M, Willaert J, Bolle L, Vanbiervliet Y, Decuypere J, Libeer F, Vandecasteele S, Peene I, Lambrecht B. Treatment of severely ill COVID-19 patients with anti-interleukin drugs (COV-AID): A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Jun 3;21(1):468. doi: 10.1186/s13063-020-04453-5. PMID 32493441

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 4th and December 6th, 2020, 342 patients were randomized. In the first randomization, 230 patients were assigned to the no IL-1 blockade group and 112 to the IL-1 blockade group, of which all received at least one dose of anakinra. In the second randomization, 115 patients were assigned to the no IL-6 blockade group, and 227 to the IL-6 blockade group, of which 114 were allocated to receive tocilizumab and 113 siltuximab.
Pre-assignment Details: 111 received siltuximab at day 1, 2 received no siltuximab due to withdrawal of consent. 113 received tocilizumab at day 1, 1 was not administered for unknown reason.
Groups:
- Anakinra: IL1-blocker: Anakinra: Anakinra will be given as a daily subcutaneous injection of 100 mg for 28 days or until hospital discharge, whichever is first
- Siltuximab: IL-6 Blocker: Siltuximab: Siltuximab will be given via single IV infusion at a dose of 11 mg/kg
- Tocilizumab: IL-6 Blocker: Tocilizumab: Tocilizumab will be given via single IV infusion at a dose of 8 mg/kg with a maximum infusion of 800 mg/injection
Period: Overall Study
Arm/Group | Usual Care | Anakinra: IL1-blocker | Siltuximab: IL-6 Blocker | Anakinra + Siltuximab | Tocilizumab: IL-6 Blocker | Anakinra + Tocilizumab
Started | 74 | 44 | 75 | 36 | 81 | 32
Randomization 1: No IL-1 Blockade | 74 | 0 | 75 | 0 | 81 | 0
Randomization 1: IL-1 Blockade | 0 | 44 | 0 | 36 | 0 | 32
Randomization 2: No IL-6 Blockade | 74 | 41 | 0 | 0 | 0 | 0
Randomization 2: IL-6 Blockade | 0 | 0 | 75 | 36 | 81 | 32
Completed | 56 | 30 | 52 | 27 | 65 | 25
Not Completed | 18 | 14 | 23 | 9 | 16 | 7
Not completed — Adverse Event | 9 | 10 | 15 | 6 | 10 | 5
Not completed — Other | 2 | 2 | 5 | 1 | 3 | 2
Not completed — Withdrawal by Subject | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 2 | 3 | 2 | 3 | 0

BASELINE CHARACTERISTICS:
Population: The study investigates IL-6 and IL-1 blockade 339 participants received IL Blockade: 227 participants IL-6 blockade + 112 participants IL-1 blockade; 345 participants No Blockade: 230 participants no IL-6 blockade + 115 participants no IL-1 blockade
Groups:
- Blockade: Patients receiving Anakinra, patients receiving Siltuximab, patients receiving Tocilizumab, patients receiving Anakinra and Siltuximab, patients receiving Anakinra and Tocilizumab
- No Blockade: Participants receiving no IL1 blockade + participants receiving no IL6 blockade
- Total: Total of all reporting groups
Arm/Group | Blockade | No Blockade | Total
Number analyzed (Participants) | 339 | 345 | 684
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: 112 participants received the IL-1 Blockade, 227 received the IL-6 Blockade, 230 received no IL-1 blockade, and 115 received no IL-6 blockade
  years
    IL-1: number analyzed (Participants) | 112 | 230 | 342
    IL-1 | 67 [56 to 74] | 64 [54 to 72] | 65 [54 to 73]
    IL-6: number analyzed (Participants) | 227 | 115 | 342
    IL-6 | 65 [54 to 73] | 64 [55 to 72] | 65 [54 to 73]
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: 112 participants received the IL-1 Blockade, 227 received the IL-6 Blockade, 230 received no IL-1 blockade, and 115 received no IL-6 blockade
  Participants
    IL-1: Female: number analyzed (Participants) | 112 | 230 | 342
    IL-1: Female | 25 | 52 | 77
    IL-1: Male: number analyzed (Participants) | 112 | 230 | 342
    IL-1: Male | 87 | 178 | 265
    IL-6: Female: number analyzed (Participants) | 227 | 115 | 342
    IL-6: Female | 52 | 25 | 77
    IL-6: Male: number analyzed (Participants) | 227 | 115 | 342
    IL-6: Male | 175 | 90 | 265
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 112 participants received the IL-1 Blockade, 227 received the IL-6 Blockade, 230 received no IL-1 blockade, and 115 received no IL-6 blockade
  Participants
    IL-1 : white: number analyzed (Participants) | 112 | 230 | 342
    IL-1 : white | 98 | 180 | 278
    IL-1: Middle Eastern-Arabian: number analyzed (Participants) | 112 | 230 | 342
    IL-1: Middle Eastern-Arabian | 11 | 29 | 40
    IL-1:Black: number analyzed (Participants) | 112 | 230 | 342
    IL-1:Black | 1 | 8 | 9
    IL-1: Asian: number analyzed (Participants) | 112 | 230 | 342
    IL-1: Asian | 1 | 6 | 7
    IL-1 : Other: number analyzed (Participants) | 112 | 230 | 342
    IL-1 : Other | 1 | 7 | 8
    IL-6 : white: number analyzed (Participants) | 227 | 115 | 342
    IL-6 : white | 184 | 94 | 278
    IL-6 : Middle Eastern-Arabian: number analyzed (Participants) | 227 | 115 | 342
    IL-6 : Middle Eastern-Arabian | 27 | 13 | 40
    IL-6: Black: number analyzed (Participants) | 227 | 115 | 342
    IL-6: Black | 8 | 1 | 9
    IL-6: Asian: number analyzed (Participants) | 227 | 115 | 342
    IL-6: Asian | 4 | 3 | 7
    IL-6: Other: number analyzed (Participants) | 227 | 115 | 342
    IL-6: Other | 4 | 4 | 8
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] — Population: BMI was available for 108 of 112 participants that received the IL-1 Blockade, for 222 of 227 participants that received the IL-6 Blockade, for 222 of 230 that received no IL-1 blockade, and for 108 of 115 participants that received no IL-6 blockade
  kg/m^2
    IL-1: number analyzed (Participants) | 108 | 222 | 330
    IL-1 | 28 [26 to 32] | 28 [26 to 32] | 28 [26 to 32]
    IL-6: number analyzed (Participants) | 222 | 108 | 330
    IL-6 | 28 [26 to 33] | 28 [26 to 31] | 28 [26 to 32]
Smoking [Count of Participants; unit: Participants] — Population: Smoking status was available for 95 of 112 participants that received the IL-1 Blockade, 181 of 227 participants that received the IL-6 Blockade, 186 of 230 participants that received no IL-1 blockade, and for 100 of 115 participants that received no IL-6 blockade
  Participants
    IL-1:No: number analyzed (Participants) | 95 | 186 | 281
    IL-1:No | 54 | 108 | 162
    IL-1: Current: number analyzed (Participants) | 95 | 186 | 281
    IL-1: Current | 7 | 11 | 18
    IL-1: Former: number analyzed (Participants) | 95 | 186 | 281
    IL-1: Former | 34 | 67 | 101
    IL-6: No: number analyzed (Participants) | 181 | 100 | 281
    IL-6: No | 101 | 61 | 162
    IL-6: Current: number analyzed (Participants) | 181 | 100 | 281
    IL-6: Current | 15 | 3 | 18
    IL-6: Former: number analyzed (Participants) | 181 | 100 | 281
    IL-6: Former | 65 | 36 | 101
Co-existing conditions [Count of Participants; unit: Participants] — Population: 112 participants received the IL-1 Blockade, 227 received the IL-6 Blockade, 230 received no IL-1 blockade, and 115 received no IL-6 blockade
  Participants
    IL-1: Arterial hypertension: number analyzed (Participants) | 112 | 230 | 342
    IL-1: Arterial hypertension | 57 | 104 | 161
    IL-1 Diabetes mellitus: number analyzed (Participants) | 112 | 230 | 342
    IL-1 Diabetes mellitus | 37 | 58 | 95
    IL-1: Cardiovascular disease: number analyzed (Participants) | 112 | 230 | 342
    IL-1: Cardiovascular disease | 29 | 41 | 70
    IL-1: Chronic kidney disease: number analyzed (Participants) | 112 | 230 | 342
    IL-1: Chronic kidney disease | 14 | 23 | 37
    IL-6: Arterial hypertension: number analyzed (Participants) | 227 | 115 | 342
    IL-6: Arterial hypertension | 115 | 46 | 161
    IL-6 Diabetes mellitus: number analyzed (Participants) | 227 | 115 | 342
    IL-6 Diabetes mellitus | 59 | 36 | 95
    IL-6: Cardiovascular disease: number analyzed (Participants) | 227 | 115 | 342
    IL-6: Cardiovascular disease | 46 | 24 | 70
    IL-6: Chronic kidney disease: number analyzed (Participants) | 227 | 115 | 342
    IL-6: Chronic kidney disease | 25 | 12 | 37
6-category ordinal scale for clinical improvement at day of randomization [Count of Participants; unit: Participants] — The 6-point ordinal scale for clinical improvement is defined as 1 = Death; 2 = Hospitalized, on invasive mechanical ventilation or ECMO; 3 = Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4 = Hospitalized, requiring supplemental oxygen; 5 = Hospitalized, not requiring supplemental oxygen; 6 = Not hospitalized. A higher score represent a better outcome Population: 112 participants received the IL-1 Blockade, 227 received the IL-6 Blockade, 230 received no IL-1 blockade, and 115 received no IL-6 blockade
  Participants
    IL-1: Hospitalized, on invasive mechanical ventilation (2): number analyzed (Participants) | 112 | 230 | 342
    IL-1: Hospitalized, on invasive mechanical ventilation (2) | 14 | 22 | 36
    IL-1: Hospitalized, on non-invasive ventilation or high flow oxygen devices (3): number analyzed (Participants) | 112 | 230 | 342
    IL-1: Hospitalized, on non-invasive ventilation or high flow oxygen devices (3) | 44 | 84 | 128
    IL-1: Hospitalized, requiring supplemental oxygen (4): number analyzed (Participants) | 112 | 230 | 342
    IL-1: Hospitalized, requiring supplemental oxygen (4) | 50 | 119 | 169
    IL-1: Hospitalized, not requiring supplemental oxygen (5): number analyzed (Participants) | 112 | 230 | 342
    IL-1: Hospitalized, not requiring supplemental oxygen (5) | 1 | 5 | 6
    IL-6: Hospitalized, on invasive mechanical ventilation (2): number analyzed (Participants) | 227 | 115 | 342
    IL-6: Hospitalized, on invasive mechanical ventilation (2) | 22 | 17 | 39
    IL-6: Hospitalized, on non-invasive ventilation or high flow oxygen devices (3): number analyzed (Participants) | 227 | 115 | 342
    IL-6: Hospitalized, on non-invasive ventilation or high flow oxygen devices (3) | 89 | 39 | 128
    IL-6: Hospitalized, requiring supplemental oxygen (4): number analyzed (Participants) | 227 | 115 | 342
    IL-6: Hospitalized, requiring supplemental oxygen (4) | 111 | 58 | 169
    IL-6: Hospitalized, not requiring supplemental oxygen (5): number analyzed (Participants) | 227 | 115 | 342
    IL-6: Hospitalized, not requiring supplemental oxygen (5) | 5 | 1 | 6
ICU at day of randomization [Count of Participants; unit: Participants] — Population: 112 participants received the IL-1 Blockade, 227 received the IL-6 Blockade, 230 received no IL-1 blockade, and 115 received no IL-6 blockade
  Participants
    IL-1: number analyzed (Participants) | 112 | 230 | 342
    IL-1 | 60 | 112 | 172
    IL-6: number analyzed (Participants) | 227 | 115 | 342
    IL-6 | 113 | 59 | 172
SOFA score at day of randomization [Median (Inter-Quartile Range); unit: units on a scale] — The Sequential Organ Failure Assessment (SOFA) Score is a mortality prediction score that is based on the degree of dysfunction of six organ systems (respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems). Score ranges from 0 (best) to 24 (worst) points. Population: SOFA score was available for 109 of 112 participants that received the IL-1 Blockade , for 208 of 227 that received the IL-6 Blockade, for 207 of 230 that received no IL-1 blockade, and for 108 of 115 that received no IL-6 blockade
  units on a scale
    IL-1: number analyzed (Participants) | 109 | 207 | 316
    IL-1 | 3 [2 to 4] | 3 [2 to 4] | 3 [2 to 4]
    IL-6: number analyzed (Participants) | 208 | 108 | 316
    IL-6 | 3 [2 to 4] | 3 [2 to 4] | 3 [2 to 4]
PaO2/FiO2 ratio at day of randomization [Median (Inter-Quartile Range); unit: ratio] — PaO2/FiO2 ratio is the ratio of the partial pressure of oxygen (PaO2) to the fraction of inspired oxygen (FiO2; PaO2/FiO2). Population: PaO2/FiO2 was available for 99 of 112 participants that received the IL-1 Blockade, for 216 of 227 participants that received the IL-6 Blockade, for 228 of 230 that received no IL-1 blockade, and for 111 of 115 participants that received no IL-6 blockade
  ratio
    IL-1: number analyzed (Participants) | 99 | 228 | 327
    IL-1 | 135 [82 to 233] | 154 [94 to 251] | 150 [90 to 248]
    IL-6: number analyzed (Participants) | 216 | 111 | 327
    IL-6 | 155 [92 to 247] | 144 [88 to 250] | 150 [90 to 248]
Vasopressor use at day of randomization [Count of Participants; unit: Participants] — Population: 112 participants received the IL-1 Blockade, 227 received the IL-6 Blockade, 230 received no IL-1 blockade, and 115 received no IL-6 blockade
  Participants
    IL-1: number analyzed (Participants) | 112 | 227 | 339
    IL-1 | 10 | 11 | 21
    IL-6: number analyzed (Participants) | 230 | 115 | 345
    IL-6 | 12 | 9 | 21
Days of symptoms at randomization [Median (Inter-Quartile Range); unit: days] — Population: Days of symptoms at randomization was available for 100 of 112 participants that received the IL-1 Blockade, for 214 of 227 participants that received the IL-6 Blockade, for 207 of 230 participants that received no IL-1 blockade, and for 107 of 115 participants that received no IL-6 blockade
  days
    IL-1: number analyzed (Participants) | 100 | 207 | 307
    IL-1 | 10 [8 to 11.5] | 10 [8 to 12] | 10 [8 to 12]
    IL-6: number analyzed (Participants) | 214 | 107 | 321
    IL-6 | 10 [8 to 12] | 10 [9 to 12] | 10 [8 to 12]
days of hospitalization at randomization [Median (Inter-Quartile Range); unit: days] — Population: 112 participants received the IL-1 Blockade, 227 received the IL-6 Blockade, 230 received no IL-1 blockade, and 115 received no IL-6 blockade
  days
    IL-1: number analyzed (Participants) | 112 | 227 | 339
    IL-1 | 3 [2 to 4] | 2 [2 to 4] | 2 [2 to 4]
    IL-6: number analyzed (Participants) | 230 | 115 | 345
    IL-6 | 3 [2 to 4] | 2 [2 to 4] | 2 [2 to 4]
Concommitant medication at day of randomization [Count of Participants; unit: Participants] — Population: 112 participants received the IL-1 Blockade, 227 received the IL-6 Blockade, 230 received no IL-1 blockade, and 115 received no IL-6 blockade
  Participants
    IL-1: Antibiotics: number analyzed (Participants) | 112 | 227 | 339
    IL-1: Antibiotics | 58 | 100 | 158
    IL-1: Remdesivir: number analyzed (Participants) | 112 | 227 | 339
    IL-1: Remdesivir | 6 | 11 | 17
    IL-1: Hydroxychloroquine: number analyzed (Participants) | 112 | 227 | 339
    IL-1: Hydroxychloroquine | 18 | 22 | 40
    IL-1: Glucocorticoids: number analyzed (Participants) | 112 | 227 | 339
    IL-1: Glucocorticoids | 72 | 141 | 213
    IL-6: Antibiotics: number analyzed (Participants) | 230 | 115 | 345
    IL-6: Antibiotics | 103 | 55 | 158
    IL-6: Remdesivir: number analyzed (Participants) | 230 | 115 | 345
    IL-6: Remdesivir | 11 | 6 | 17
    IL-6: Hydroxychloroquine: number analyzed (Participants) | 230 | 115 | 345
    IL-6: Hydroxychloroquine | 25 | 15 | 40
    IL-6: Glucocorticoids: number analyzed (Participants) | 230 | 115 | 345
    IL-6: Glucocorticoids | 141 | 72 | 213
CRP at day of randomization [Median (Inter-Quartile Range); unit: mg/mL] — Population: CRP was available for all 112 participants that received the IL-1 Blockade, for 226 of 227 participants that received the IL-6 Blockade, for 224 of 230 that received no IL-1 blockade, and for 114 of 115 participants that received no IL-6 blockade
  mg/mL
    IL-1: number analyzed (Participants) | 112 | 224 | 336
    IL-1 | 148 [86 to 211] | 123 [81 to 183] | 129 [83 to 197]
    IL-6: number analyzed (Participants) | 226 | 114 | 340
    IL-6 | 129 [83 to 193] | 129 [81 to 199] | 129 [83 to 197]
Lymphocyte count at day of randomization [Median (Inter-Quartile Range); unit: 10^3 cells /µL] — Population: Lymphocyte count at day of randomization was available for 108 of 112 participants that received the IL-1 Blockade, for 220 of 227 participants that received the IL-6 Blockade, for 224 of 230 that received no IL-1 blockade, and for 112 of 115 participants that received no IL-6 blockade
  10^3 cells /µL
    IL-1: number analyzed (Participants) | 108 | 224 | 332
    IL-1 | 0.7 [0.5 to 0.9] | 0.7 [0.5 to 0.9] | 0.7 [0.5 to 0.9]
    IL-6: number analyzed (Participants) | 220 | 112 | 332
    IL-6 | 0.6 [0.5 to 0.9] | 0.7 [0.5 to 0.9] | 0.7 [0.5 to 0.9]
Ferritin at day of randomization [Median (Inter-Quartile Range); unit: µg/L] — Population: Ferritin at day of randomization was available for 109 of 112 participants that received the IL-1 Blockade, for 222 of 227 participants that received the IL-6 Blockade, for 223 of 230 that received no IL-1 blockade, and for 110 of 115 participants that received no IL-6 blockade
  µg/L
    IL-1: number analyzed (Participants) | 109 | 223 | 332
    IL-1 | 1672 [1187 to 2509] | 1688 [1166 to 2811] | 1687 [1173 to 2725]
    IL-6: number analyzed (Participants) | 222 | 110 | 332
    IL-6 | 1680 [1149 to 2759] | 1749 [1205 to 2619] | 1687 [1173 to 2725]
D-dimers at day of randomization [Median (Inter-Quartile Range); unit: ng/mL] — Population: D-dimers at day of randomization was available for 90 of 112 participants that received the IL-1 Blockade, for 192 of 227 participants that received the IL-6 Blockade, for 193 of 230 that received no IL-1 blockade, and for 91 of 115 participants that received no IL-6 blockade
  ng/mL
    IL-1: number analyzed (Participants) | 90 | 193 | 283
    IL-1 | 1091 [510 to 1847] | 1000 [560 to 1490] | 1011 [551 to 1688]
    IL-6: number analyzed (Participants) | 192 | 91 | 283
    IL-6 | 1000 [550 to 1600] | 1099 [567 to 1780] | 1011 [551 to 1688]
LDH at day of randomization [Median (Inter-Quartile Range); unit: IU/L] — Population: LDH was available for 111 of 112 participants that received the IL-1 Blockade, for 224 of 227 participants that received the IL-6 Blockade, for 224 of 230 that received no IL-1 blockade, and for 111 of 115 participants that received no IL-6 blockade
  IU/L
    IL-1: number analyzed (Participants) | 111 | 224 | 335
    IL-1 | 445 [356 to 537] | 430 [356 to 559] | 435 [356 to 543]
    IL-6: number analyzed (Participants) | 224 | 111 | 335
    IL-6 | 435 [356 to 511] | 435 [356 to 589] | 435 [356 to 543]
IL-1-RA at day of randomization [Median (Inter-Quartile Range); unit: ng/mL] — Population: IL-1-RA at day of randomization was available for 108 of 112 participants that received the IL-1 Blockade, for 216 of 227 participants that received the IL-6 Blockade, for 216 of 230 that received no IL-1 blockade, and for 108 of 115 participants that received no IL-6 blockade
  ng/mL
    IL-1: number analyzed (Participants) | 108 | 216 | 324
    IL-1 | 940 [527 to 1631] | 903 [525 to 2150] | 916 [525 to 1977]
    IL-6: number analyzed (Participants) | 216 | 108 | 324
    IL-6 | 931 [513 to 1976] | 885 [531 to 1978] | 916 [525 to 1977]
IL-1B at day of randomization [Median (Inter-Quartile Range); unit: fg/mL] — Population: IL-1B at day of randomization was available for 104 of 112 participants that received the IL-1 Blockade, for 213 of 227 participants that received the IL-6 Blockade, for 210 of 230 that received no IL-1 blockade, and for 107 of 115 participants that received no IL-6 blockade
  fg/mL
    IL-1: number analyzed (Participants) | 104 | 213 | 317
    IL-1 | 44 [11 to 99] | 60 [22 to 127] | 56 [19 to 117]
    IL-6: number analyzed (Participants) | 210 | 107 | 317
    IL-6 | 52 [18 to 99] | 74 [20 to 131] | 56 [19 to 117]
IL-6 at day of randomization [Median (Inter-Quartile Range); unit: pg/mL] — Population: IL-6 at day of randomization was available for 108 of 112 participants that received the IL-1 Blockade, for 216 of 227 participants that received the IL-6 Blockade, for 216 of 230 that received no IL-1 blockade, and for 108 of 115 participants that received no IL-6 blockade
  pg/mL
    IL-1: number analyzed (Participants) | 108 | 216 | 324
    IL-1 | 8 [3 to 20] | 10 [3 to 23] | 9 [3 to 21]
    IL-6: number analyzed (Participants) | 216 | 108 | 324
    IL-6 | 9 [3 to 24] | 8 [3 to 20] | 9 [3 to 21]

OUTCOME MEASURES:

1. Primary Outcome: Time to Clinical Improvement
Description: Time to Clinical Improvement is defined as the time from randomization to either an increase of at least two points on a six category ordinal scale from the status at randomization or live discharge from the hospital.The 6-point ordinal scale for clinical improvement is defined as 1 = Death; 2 = Hospitalized, on invasive mechanical ventilation or ECMO; 3 = Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4 = Hospitalized, requiring supplemental oxygen; 5 = Hospitalized, not requiring supplemental oxygen; 6 = Not hospitalized. A higher score represent a better outcome
Time Frame: at day 15
Population: Participants were re-grouped and analyzed based on the following pre-specified factorial combinations: IL-1 Blockade, No IL-1 Blockade, IL-6 Blockade, No IL-6 Blockade
Measure: Median (95% Confidence Interval); unit: days
Groups:
- IL 1 Blockade: All patients received Kineret® (Anakinra) 100mg pre-filled syringe given 1x / day for 28 days (or until discharge from hospital). Some patients also received Sylvant® (Siltuximab) single IV infusion from 100mg powder concentrate and 400mg powder concentrate, OR Roactemra® (tocilizumab) IV- Infusion prepared starting from flasks containing 400mg/20ml stock solution (to dilute for infusion) or from Prefilled syringe 162mg / 0.9ml SC
- No IL-1 Blockade: Some patients received IL-6 blockade with Sylvant® (Siltuximab) single IV infusion from 100mg powder concentrate and 400mg powder concentrate, OR Roactemra® (tocilizumab) IV- Infusion prepared starting from flasks containing 400mg/20ml stock solution (to dilute for infusion) or from Prefilled syringe 162mg / 0.9ml SC
- IL-6 Blockade: Patients received either Sylvant® (Siltuximab) single IV infusion from 100mg powder concentrate and 400mg powder concentrate, OR Roactemra® (tocilizumab) IV- Infusion prepared starting from flasks containing 400mg/20ml stock solution (to dilute for infusion) or from Prefilled syringe 162mg / 0.9ml SC Some patients also received Kineret® (Anakinra) 100mg pre-filled syringe given 1x / day for 28 days (or until discharge from hospital)
- No IL-6 Blockade: Some patients received Kineret® (Anakinra) 100mg pre-filled syringe given 1x / day for 28 days (or until discharge from hospital)
Arm/Group | IL 1 Blockade | No IL-1 Blockade | IL-6 Blockade | No IL-6 Blockade
Number analyzed (Participants) | 112 | 230 | 227 | 115
days | 12 [10 to 16] | 12 [10 to 15] | 11 [10 to 16] | 12 [11 to 16]

2. Secondary Outcome: Time Untill Discharge
Time Frame: during hospital admission (up to 28 days)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | IL 1 Blockade | No IL-1 Blockade | IL-6 Blockade | No IL-6 Blockade
Number analyzed (Participants) | 112 | 230 | 227 | 115
days | 14 [11 to 19] | 12 [11 to 18] | 12 [11 to 18] | 13 [11 to 19]

3. Secondary Outcome: Time Until Independence From Supplemental Oxygen or Discharge
Time Frame: during hospital admission (up to 28 days)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | IL 1 Blockade | No IL-1 Blockade | IL-6 Blockade | No IL-6 Blockade
Number analyzed (Participants) | 112 | 230 | 227 | 115
days | 12 [10 to 20] | 12 [10 to 15] | 11 [10 to 15] | 12 [10 to 15]

4. Secondary Outcome: Time Until Independence From Invasive Ventilation
Time Frame: during hospital admission (up to 54 days)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | IL 1 Blockade | No IL-1 Blockade | IL-6 Blockade | No IL-6 Blockade
Number analyzed (Participants) | 112 | 230 | 227 | 115
days | 21 [8 to NA] — Upper limit of 95% CI not estimable due to insufficient numbers of participants who reached independence of invasive mechanical ventilation | 27 [9 to NA] — Upper limit of 95% CI not estimable due to insufficient numbers of participants who reached independence of invasive mechanical ventilation | 23 [8 to NA] — Upper limit of 95% CI not estimable due to insufficient numbers of participants who reached independence of invasive mechanical ventilation | 54 [9 to NA] — Upper limit of 95% CI not estimable due to insufficient numbers of participants who reached independence of invasive mechanical ventilation

5. Secondary Outcome: Number of Days in ICU
Time Frame: during hospital admission (up to 28 days)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | IL 1 Blockade | No IL-1 Blockade | IL-6 Blockade | No IL-6 Blockade
Number analyzed (Participants) | 112 | 230 | 227 | 115
days | 11 [8 to 15] | 10 [8 to 13] | 11 [8 to 14] | 10 [7 to 15]

6. Secondary Outcome: Number of Days in ICU in Patients Ventilated at Day of Randomization
Time Frame: during hospital admission (up to 28 days)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | IL 1 Blockade | No IL-1 Blockade | IL-6 Blockade | No IL-6 Blockade
Number analyzed (Participants) | 112 | 230 | 227 | 115
days | 20 [15 to 27] | 22 [17 to 29] | 20 [16 to 27] | 22 [16 to 29]

7. Secondary Outcome: Number of Days Without Supplemental Oxygen Use
Time Frame: during hospital admission (up to 28 days)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | IL 1 Blockade | No IL-1 Blockade | IL-6 Blockade | No IL-6 Blockade
Number analyzed (Participants) | 112 | 230 | 227 | 115
days | 9 [7 to 12] | 9 [7 to 11] | 10 [8 to 12] | 8 [6 to 11]

8. Secondary Outcome: Number of Invasive Ventilator Days
Time Frame: during hospital admission (up to 28 days)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | IL 1 Blockade | No IL-1 Blockade | IL-6 Blockade | No IL-6 Blockade
Number analyzed (Participants) | 112 | 230 | 227 | 115
days | 5 [3 to 9] | 5 [3 to 7] | 5 [3 to 7] | 5 [3 to 9]

9. Secondary Outcome: Number of Invasive Ventilator Days in Patients Ventilated at Day of Randomization
Time Frame: during hospital admission (up to 28 days)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | IL 1 Blockade | No IL-1 Blockade | IL-6 Blockade | No IL-6 Blockade
Number analyzed (Participants) | 112 | 230 | 227 | 115
days | 15 [11 to 20] | 16 [13 to 21] | 15 [12 to 20] | 16 [12 to 22]

10. Secondary Outcome: Number of Invasive Ventilator-free Days
Time Frame: during hospital admission (up to 28 days)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | IL 1 Blockade | No IL-1 Blockade | IL-6 Blockade | No IL-6 Blockade
Number analyzed (Participants) | 112 | 230 | 227 | 115
days | 18 [15 to 21] | 18 [16 to 20] | 18 [17 to 20] | 17 [15 to 20]

11. Secondary Outcome: Number of Invasive Ventilator-free Days in Patients Ventilated at Day of Randomization
Time Frame: during hospital admission (up to 28 days)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | IL 1 Blockade | No IL-1 Blockade | IL-6 Blockade | No IL-6 Blockade
Number analyzed (Participants) | 112 | 230 | 227 | 115
days | 6 [3 to 14] | 6 [3 to 13] | 7 [4 to 15] | 5 [2 to 12]

12. Secondary Outcome: Percentage of Days in ICU
Description: Number of days the participants were ventilated, relative to the number of days participants were alive during the first 28 days after randomization. This was calculated as the number of days with need for invasive ventilation / number of days alive during first 28 days, multiplied by 100 (to obtain a percentage).
Time Frame: first 28 days after randomization
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: percentage of days
Arm/Group | IL 1 Blockade | No IL-1 Blockade | IL-6 Blockade | No IL-6 Blockade
Number analyzed (Participants) | 112 | 230 | 227 | 115
percentage of days | 42 [31 to 56] | 36 [29 to 46] | 38 [30 to 48] | 40 [29 to 54]

13. Secondary Outcome: Percentage of Invasive Ventilator Days
Description: Number of days the participant spent in the ICU, relative to the number of days the patient was alive during the first 28 days after randomization. This was calculated as the number of days in ICU during first 28 days / number of days alive during first 28 days, multiplied by 100 (to obtain a percentage).
Time Frame: the first 28 days after randomization
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: percentage of days
Arm/Group | IL 1 Blockade | No IL-1 Blockade | IL-6 Blockade | No IL-6 Blockade
Number analyzed (Participants) | 112 | 230 | 227 | 115
percentage of days | 23 [14 to 38] | 21 [14 to 31] | 21 [14 to 30] | 23 [14 to 38]

14. Secondary Outcome: Time Until First Use of High-flow Oxygen Device, Ventilation, or Death
Time Frame: during hospital admission (up to 28 days)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | IL 1 Blockade | No IL-1 Blockade | IL-6 Blockade | No IL-6 Blockade
Number analyzed (Participants) | 112 | 230 | 227 | 115
days | NA [NA to NA] — < 50% reached event | NA [NA to NA] — < 50% reached event | NA [NA to NA] — < 50% reached event | NA [NA to NA] — < 50% reached event

ADVERSE EVENTS:
Time Frame: AE's are recorded from randomisation until the end of the study, 5 months
Arm/Group | Usual Care | Anakinra | Siltuximab | Anakinra + Siltuximab | Tocilizumab | Anakinra + Tocilizumab
All-Cause Mortality (participants affected / at risk) | 9/74 | 10/44 | 15/75 | 6/36 | 10/81 | 5/32
Serious Adverse Events (participants affected / at risk) | 14/74 | 12/44 | 21/75 | 8/36 | 15/81 | 9/32
Other Adverse Events (participants affected / at risk) | 37/74 | 25/44 | 15/75 | 17/36 | 35/81 | 17/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=74) | Anakinra (N=44) | Siltuximab (N=75) | Anakinra + Siltuximab (N=36) | Tocilizumab (N=81) | Anakinra + Tocilizumab (N=32)
Arterial thromboembolism (Vascular disorders) | 0 | 0 | 21 | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0
Other (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
Anaphylaxis (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 3 | 2 | 0 | 0 | 2 | 1
postoperative haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Asystole (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 1 | 0 | 1 | 0
Other (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Mitral valve disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 9 | 2 | 6 | 1
Other (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Edema cerebral (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Intracranial haemorrhage (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Jejunal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hepatic infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 2
Sepsis (Infections and infestations) | 3 | 5 | 6 | 3 | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=74) | Anakinra (N=44) | Siltuximab (N=75) | Anakinra + Siltuximab (N=36) | Tocilizumab (N=81) | Anakinra + Tocilizumab (N=32)
Hypertension (Vascular disorders) | 4 | 3 | 4 | 1 | 3 | 3
Hypotension (Vascular disorders) | 4 | 3 | 1 | 0 | 1 | 1
Thromboembolic event (Vascular disorders) | 1 | 3 | 4 | 0 | 3 | 0
Alanine aminotransferase increased (Investigations) | 3 | 3 | 7 | 3 | 7 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 2 | 5 | 2 | 5 | 0
Creatinine increased (Investigations) | 2 | 0 | 1 | 2 | 0 | 0
GGT increased (Investigations) | 2 | 2 | 5 | 0 | 2 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 2
Platelet count decreased (Investigations) | 0 | 0 | 4 | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 3 | 0 | 7 | 1 | 0 | 3
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 8 | 2 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 1 | 2
Other (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 2 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 3 | 4 | 3 | 2 | 0
Other (Blood and lymphatic system disorders) | 0 | 3 | 4 | 4 | 3 | 0
Delirium (Psychiatric disorders) | 3 | 2 | 4 | 0 | 2 | 1
Constipation (Gastrointestinal disorders) | 10 | 5 | 9 | 4 | 8 | 7
Diarrhoea (Psychiatric disorders) | 2 | 3 | 3 | 1 | 2 | 1
Gastroparesis (Psychiatric disorders) | 3 | 3 | 1 | 0 | 3 | 1
Nausea (Gastrointestinal disorders) | 4 | 0 | 2 | 2 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 3 | 2 | 0 | 1 | 0
Other (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 2
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 — lower limb
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 4 | 1 | 2 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 4 | 0 | 3 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 2 | 3 | 2 | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 1 | 0 | 1
Other (Metabolism and nutrition disorders) | 2 | 1 | 5 | 1 | 0 | 2
Bacteraemia (Infections and infestations) | 2 | 2 | 2 | 0 | 0 | 2
Lung infection (Infections and infestations) | 7 | 4 | 8 | 3 | 8 | 5
Sepsis (Infections and infestations) | 3 | 0 | 5 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 4 | 1 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/38/NCT04330638/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/38/NCT04330638/SAP_001.pdf